CLINICAL TRIAL: NCT01768533
Title: Pediatric Behavioral Informatics to Prevent Cancer
Acronym: TIDE
Status: Completed | Type: Observational
Sponsor: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Julie Wright, Assistant Professor, University of Massachusetts, Boston
Other Study IDs: 5K07CA113643 (NIH)
Record Dates: First submitted 2012-12-26; First posted 2013-01-15 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Obesity
Keywords: pediatric; obesity; prevention; health behaviors; guidelines
MeSH Terms: conditions — Obesity; Health Behavior

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey: A lifestyle survey was administered to primary-care givers or legal guardians who take their children 4-10 y/o to the pediatric well-child visits.

SUMMARY:
The goal of this study is to do formative research which will lead ultimately to the development of a computer-based system called Tailored Information for Diet and Exercise or TIDE for short. TIDE will target energy balance behaviors to prevent the onset of obesity in children. The system will be used by physicians and parents/primary care givers in pediatric primary care practices with the aim of improving parent-pediatrician interactions related to counseling and anticipatory guidance on energy balance behaviors. The aim of this study is to develop a one-two page, paper-pencil proxy questionnaire that is used to query the parent of the child in the waiting room and assesses topic areas related to energy balance behaviors (EBB). The questionnaire will be referred to as the energy balance behaviors questionnaire (EBB-Q). This will require focus groups, cognitive testing of the questionnaire, and survey administration.

ELIGIBILITY:
Inclusion Criteria:

* primary care givers or legal guardians of children 4-10 years of age who has attended the last two well-child visits with their child

Exclusion Criteria:

* parent cares for a child who is on a special diet prescribed by pediatrician

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General population of parents with children ages 4-10 years who reside in the Greater Boston area. Parents are defined as primary care givers or legal guardians who take primary responsibility for the child's health which includes attending the child's well-care visits.
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
sugar-sweetened beverages | one time point (baseline only)
  Behavioral outcome measure of the amount of sugar-sweetened beverages consumed.

SECONDARY OUTCOMES:
BMI | one time point (baseline only)
  weight status as defined by body mass index (BMI)

OTHER OUTCOMES:
Physical activity | one time point (baseline only)
  amount of time spent in moderate or greater physical activity
fruit and vegetables | one time point (baseline only)
  amount of fruit servings and vegetable servings consumed per day.
screen time | one time point (baseline only)
  amount of time spent watching television or recreational videos or computers

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Wright, PhD, Principal Investigator — UMass Boston
Locations (1):
- UMass Boston, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Wright JA, Whiteley JA, Watson BL, Sheinfeld Gorin SN, Hayman LL. Tailored communications for obesity prevention in pediatric primary care: a feasibility study. Health Educ Res. 2018 Feb 1;33(1):14-25. doi: 10.1093/her/cyx063. PMID 29112721
- [Derived] Wright JA, Adams WG, Laforge RG, Berry D, Friedman RH. Assessing parental self-efficacy for obesity prevention related behaviors. Int J Behav Nutr Phys Act. 2014 Apr 22;11:53. doi: 10.1186/1479-5868-11-53. PMID 24750693